CLINICAL TRIAL: NCT06124079
Title: The Implementation of a Post-operative Communication App to Improve Pain Control and Opioid Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SURG-2023-32217
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Placebo Comparator): Standard care currently consists of education materials with the after visit summary (available in MyChart) around opioid use and precautions and disposal information.
  Interventions: Other: Standard care
- Interactive messaging service (Experimental): Participants will be randomized to one of 2 specific versions of OPY.
  Interventions: Other: OPY interactive messaging service

INTERVENTIONS:
Other: OPY interactive messaging service — 2 specific versions of OPY. information. Each version will deliver the same instructions and information about pain management recommendations, and collect the same information about patient pain experience and side effects. The two versions differ in the motivational techniques interspersed throughout the OPY experience.
  Arms: Interactive messaging service
Other: Standard care — Standard care currently consists of education materials with the after visit summary (available in MyChart) around opioid use and precautions and disposal information.
  Arms: standard care

SUMMARY:
Digital communication tools are becoming ubiquitous in healthcare, though their impact on patient/provider communication, healthcare utilization, and outcomes remains poorly established. M Health Fairview (MHFV) in collaboration with the Center for Learning Health System Sciences (CLHSS) Rapid Eval team will be evaluating one such communication application: OPY, which leverages the Epic-Care Companion functionality to remove barriers in communicating with the patient's care team. This project will evaluate the effectiveness of a digital, post-operative patient engagement tool (Epic-Care Companion made available through MyChart), OPY, which has the goal of preventing patients from becoming addicted to opioids or to suffer from opioid misuse or diversion. In the proposed pragmatic trial, standard care with education available in MyChart and the patient after visit summary will be augmented by OPY. OPY is available to patients starting the same day they go home from surgery with a new opioid prescription. OPY provides a daily interactive experience that collects patient pain and side-effect information, provides advice for pain management, and uses behavioral "nudges" to encourage timely weaning and responsible disposal of opioid medications. The primary goal of this project is to evaluate the effect of two versions of OPY on measures of opiate use relative to the standard of care in a pragmatic randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Surgery at The M Health Fairview Clinics and Surgery Center - Maple Grove (Maple Grove) or M Health Fairview Clinics and Surgery Center - Minneapolis (CSC)

  ▪ Currently, only outpatient surgeries are performed at CSC and Maple Grove
* Active opioid prescription (prescribed between 30 days prior to surgery, until day of surgery)
* Patient class (outpatient or same day surgery)
* Never previously randomized or exposed to OPY

Exclusion Criteria:

* Age < 18
* Chronic opiate use defined as:

  * Patients aged 18 and older and
  * 3 or more opioid dispensing events, in the last 12 months with at least 1 of these events in the last 6 months.
* Any long acting opioid prescription in the last 6 months
* Interpreter needed - YES selected (EPT840)
* Patient has a Health Proxy (Legal Guardian) designated in Epic
* Patients who have opted out of clinical research
* Patients with an active palliative care referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Opiate use at 14 days | 14 days
  Opiate use at 14 days is defined as any active opioid script on day 14 post surgery. This information will be collected from the electronic health record.

SECONDARY OUTCOMES:
Number of days between initiation of opioid therapy and opioid-free pain control | 24 months
Interval time between opioid doses | 24 months
Daily pain scores | 24 months
Number and cause of patient initiated outreach events | 24 months
  from the care companion app
Number of MyChart messages | 30 days post-op
Number of Phone notes | 30 days post-op
90-day Hospitalization Rates | 90 days
Hospital length of stay | 24 months
Repeat Surgery Rates | 24 months
Outpatient encounter Rates | 24 months
Referral rates | 24 months
completion of referral of pain management rates | 24 months
Opiate use rates | 90 and 120 days
OPY utilization | 1,3,7, 14, and 30 days
all-cause mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Melton-Meaux, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Rizvi RF, Schoephoerster JA, Desphande SS, Usher M, Oien AE, Peters MM, Loth MS, Bahr MW, Ventz S, Koopmeiners JS, Melton GB. Decreasing Opioid Addiction and Diversion Using Behavioral Economics Applied Through a Digital Engagement Solution: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 8;13:e52882. doi: 10.2196/52882. PMID 38457203